CLINICAL TRIAL: NCT00617539
Title: A Phase II Study of Irinotecan and Temozolomide in Breast Cancer Patients With Brian Metastases That Have Progressed After Stereotactic Radiosurgery or Whole Brain Radiation
Brief Title: Irinotecan and Temozolomide in Treating Patients With Breast Cancer Who Have Received Previous Treatment for Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05751; UCSF-05751
Record Dates: First submitted 2008-02-15; First posted 2008-02-18 (Estimated); Results first posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer; Metastatic Cancer
Keywords: recurrent breast cancer; stage IV breast cancer; male breast cancer; tumors metastatic to brain
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Breast Neoplasms, Male; Brain Neoplasms | interventions — Irinotecan; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- irinotecan and temozolomide (Experimental)
  Interventions: Drug: irinotecan hydrochloride; Drug: temozolomide

INTERVENTIONS:
Drug: irinotecan hydrochloride
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan and temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects of giving irinotecan together with temozolomide and to see how well it works in treating patients with breast cancer who have received previous treatment for brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the objective response rate systemically and in the CNS to the combination of irinotecan hydrochloride and temozolomide among patients with breast cancer and progressive brain metastases that have progressed after previous treatment for brain metastases.
* To determine the toxicities associated with the combination of irinotecan hydrochloride and temozolomide in breast cancer patients with progressive brain metastases.

Secondary

* To evaluate the time to first progression at any site (CNS or extra-CNS) in patients treated with the combination of irinotecan hydrochloride and temozolomide.
* To evaluate the overall survival of patients treated with the combination of irinotecan hydrochloride and temozolomide for brain metastases.

OUTLINE: Patients receive irinotecan IV on days 1 and 15 and oral temozolomide on days 1-7 and 15-21. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 4 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer with radiographically confirmed metastases to the brain

  * Extracranial metastases allowed
* Must have demonstrated progression of brain metastases after prior treatment for brain metastases, including any of the following:

  * External beam radiotherapy
  * Brachytherapy
  * Stereotactic radiosurgery
  * Surgery
  * Chemotherapy
  * Treatments with investigational drugs, biologics, or devices
* Disease progression in the CNS must meet ≥ 1 of the following criteria:

  * New lesions in the CNS on an imaging study (contrast-enhanced CT scan or MRI)
  * Progressive lesions on an imaging study (contrast-enhanced CT scan or MRI)
* New or progressive lesions that do not meet measurable disease definition allowed
* Leptomeningeal disease allowed if concurrent progression or parenchymal brain metastases
* Not a candidate for surgical resection and/or further stereotactic radiosurgery
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* ECOG performance status 0-2
* Life expectancy ≥ 1 month
* Hemoglobin ≥ 10 g/dL (transfusion allowed)
* ANC ≥ 1,500/mm³
* Granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 mg/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 3 times ULN
* Must be able to swallow and retain oral medications
* No other active malignancy except for any of the following:

  * Curatively treated basal or squamous cell carcinoma of the skin
  * Carcinoma in situ of the cervix
  * Other malignancies considered disease-free
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of immediate or delayed-type hypersensitivity reaction to gadolinium contrast agents or other contraindication to gadolinium contrast
* No other known contraindication to MRI including, but not limited to, any of the following:

  * Cardiac pacemaker
  * Implanted cardiac defibrillator
  * Brain aneurysm clips
  * Cochlear implant
  * Ocular foreign body
  * Shrapnel
* No active or uncontrolled infection

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from the side effects of prior chemotherapy, surgery, or radiotherapy for extracranial disease or brain metastases
* Concurrent trastuzumab, bisphosphonate, and/or corticosteroid therapy allowed
* At least 1 week since prior or on current stable dose of corticosteroid therapy
* Patients on an enzyme-inducing anti-epileptic agent (EIAE) or valproic acid are eligible if they are switched to an alternate non-EIAE medication
* Concurrent coumadin allowed
* No prophylactic use of filgrastim (G-CSF) during first course of treatment

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-02; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Melisko, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Irinotecan and Temozolomide: 125 mg/m^2 irinotecan hydrochloride administered intravenously on days 1 and 15 of a 28 day cycle
  100 mg/m^2 temozolomide orally for seven days on days 1-7 and days 15-21 of a 28 day cycle
Period: Overall Study
Arm/Group | Irinotecan and Temozolomide
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Irinotecan and Temozolomide
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 53.5 [31 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Objective Treatment Response (Complete or Partial) in the CNS
Description: Imaging was performed at 8-week intervals to assess response to treatment. Patients with known or suspected leptomeningeal disease were deemed to have a complete response if CSF cytology converted to negative (if positive at baseline) and all meningeal enhancement or nodularity of brain and/or spine MRI resolved. A modified RECIST 1.0 criteria was used to assess CNS response for patients with new or progressing brain metastases. In this modified RECIST criteria, CNS lesions <1cm were not considered measurable, but were considered evaluable for response and progression. Progressive disease for patients with lesions <1 cm was defined as follows: growth of a lesion from less than or equal to 5 mm to greater than or equal to 10mm; or, growth of a 6-9 mm lesion by at least 5 mm in the case of non-target parenchymal brain metastases.
Time Frame: Baseline scan prior to study entry was performed within 14 days of cycle 1 day 1, then every 8 weeks from then until disease progression or up to 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Irinotecan and Temozolomide: irinotecan hydrochloride administered intravenously (IV) at a starting dose of 125 mg/m2 on days 1 and 15 of a 28 day cycle
  temozolomide orally for seven days at a starting dose of 100 mg/m2 on days 1-7 and days 15-21 of a 28 day cycle
Arm/Group | Irinotecan and Temozolomide
Number analyzed (Participants) | 30
Participants | 2

2. Secondary Outcome: Time to First Progression in CNS
Description: Imaging at 8-week intervals to assess response to treatment. A modified RECIST 1.0 criteria was used to assess response and time to progression in the CNS for patients with progressing brain metastases. In this modified RECIST criteria, CNS lesions <1cm were not considered measurable, but were considered evaluable for response and progression. Progressive disease for patients with lesions <1 cm was defined as follows: growth of a lesion from less than or equal to 5 mm to greater than or equal to 10mm; or, growth of a 6-9 mm lesion by at least 5 mm in the case of non-target parenchymal brain metastases.
  If patient did not come back for a follow up scan after clinical deterioration, patient was only considered stable up to the time of the last scan per protocol and time to progression would be from cycle 1 day 1 to the last scan they completed that was stable.
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: Days
Arm/Group | Irinotecan and Temozolomide
Number analyzed (Participants) | 30
Days | 70 [13 to 444]

3. Secondary Outcome: Overall Time of Survival
Description: Time from initiation of study participation until death
Time Frame: Time from initiation of study participation until death or up to 3 years
Measure: Median (Full Range); unit: Days
Arm/Group | Irinotecan and Temozolomide
Number analyzed (Participants) | 30
Days | 146 [20 to 1043]

4. Secondary Outcome: Number of Patients Whose Circulating Tumor Cells (CTCs) Decreased From >5 to <5 CTCs Per 7.5 mL
Description: CTCs were measured in blood using the Cellsearch(R) assay in 14 of the 20 patients measured at baseline
Time Frame: CTCs drawn on cycle 1 day 1, collection at 8 week intervals on patients who did not progress on their 8 week scans up to 2 years
Population: Of 20 patients with CTCs measured at baseline, 14 were also measured at 8 weeks
Measure: Number; unit: participants
Groups:
- Irinotecan and Temozolomide: irinotecan hydrochloride administered intravenously at a starting dose of 125 mg/m2 on days 1 and 15 of a 28 day cycle
  temozolomide orally for seven days at a starting dose of 100 mg/m2 on days 1-7 and days 15-21 of a 28 day cycle
Arm/Group | Irinotecan and Temozolomide
Number analyzed (Participants) | 14
participants | 1

5. Primary Outcome: Number of Patients Experiencing a Clinical Benefit
Description: The number of patients experiencing a clinical benefit is the sum of patients with an objective response plus patients with stable disease at ≥ 16 weeks from cycle 1 day 1 (first day of treatment). If a patient did not come back for a follow up scan after clinical deterioration, then they were only considered stable up to the time of the last scan they had per protocol.
Time Frame: From 1 day 1 (first day of treatment) every 8 weeks until scan shows disease progression or up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Irinotecan and Temozolomide
Number analyzed (Participants) | 30
Participants | 7

ADVERSE EVENTS:
Time Frame: During study treatment (up to 3 years)
Description: Only one mortality during study treatment window. All other mortalities occured during the long term follow up and are not reported in the All-Cause Mortality module.
Groups:
- Irinotecan and Temozolomide: irinotecan hydrochloride administered intravenously at a starting dose of 125 mg/m2 on days 1 and 15 of a 28 day cycle, and temozolomide orally for seven days at a starting dose of 100 mg/m2 on days 1-7 and days 15-21 every 28 days.
Arm/Group | Irinotecan and Temozolomide
All-Cause Mortality (participants affected / at risk) | 14/30
Serious Adverse Events (participants affected / at risk) | 16/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Irinotecan and Temozolomide (N=30)
Infection (Infections and infestations) | 4
Hyponatremia (Renal and urinary disorders) | 4
Fatigue (General disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Transaminitis (Hepatobiliary disorders) | 1
Neuropathy (Nervous system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 16
Leukopenia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 5
Anemia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Dehydration (General disorders) | 2
Alkaline phosphatase increased (General disorders) | 1
Mental status change (Nervous system disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Weakness (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Irinotecan and Temozolomide (N=30)
Infection (Infections and infestations) | 5
Hyponatremia (Renal and urinary disorders) | 1
Fatigue (General disorders) | 15
Vomiting (Gastrointestinal disorders) | 15
Nausea (Gastrointestinal disorders) | 22
Diarrhea (Gastrointestinal disorders) | 15
Transaminitis (Hepatobiliary disorders) | 5
Neuropathy (Nervous system disorders) | 7
Hypocalcemia (Endocrine disorders) | 8
Mucositis (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 8
Hypokalemia (Renal and urinary disorders) | 6
Anorexia (General disorders) | 6
Dizziness (Nervous system disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 9
Dyspepsia (Gastrointestinal disorders) | 6
Lymphopenia (Blood and lymphatic system disorders) | 5
Leukopenia (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 8
Anemia (Blood and lymphatic system disorders) | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Dehydration (General disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Fever (General disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 3
Hyperbilirubinemia (Hepatobiliary disorders) | 3
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 2
Weakness (General disorders) | 2
Xerostomia (Gastrointestinal disorders) | 2
Abdominal pain (General disorders) | 1
Bruising (Blood and lymphatic system disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Hypomagnesemia (General disorders) | 1
Creatinine increased (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes